CLINICAL TRIAL: NCT05757830
Title: Metabolic Consumption, Cardiorespiratory Effort, Cardiac Autonomic Control and Fatigability During Exoskeleton-assisted (the U&O Suite) sit-to Stand Maneuver and Walking in People With Neurological Diseases With Moderate to Severe Gait Disability.
Brief Title: PURO - PUlmonary Rehabilitation With O-RAGT Platform
Acronym: PURO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Roessingh Research and Development (Other); Hospital Nacional de Parapléjicos de Toledo (Other); Lithuanian University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 825003
Record Dates: First submitted 2023-01-19; First posted 2023-03-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis; Spinal Cord Injury; Stroke; Traumatic Brain Damage
MeSH Terms: conditions — Multiple Sclerosis; Spinal Cord Injuries; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exoskeleton-assisted arm (Experimental): Each subject will perform 3 experimental conditions with and without the exoskeleton to assess the impact of exoskeleton assisted walking on metabolic consumption and cardiorespiratory effort compared to conventional overground walking training without an exoskeleton
  Interventions: Device: UANGO suite exoskeleton

INTERVENTIONS:
Device: UANGO suite exoskeleton — Each subject will perform 3 experimental conditions (Condition 1: Walking without exoskeleton; Condition 2: Walking with exoskeleton; Condition 3: Walking with exoskeleton and walker).
  Each condition includes 5 triasl (Trial 1 - Sitting: 5 minutes, sitting at rest in comfortable position; Trial 2 - Standing: 5 minutes, with assistance; Trial 3 - Comfortable speed Walking (100% assisted): 4 min during back-and-forth locomotion on a 20-m length linear flat path; Trial 4 - Comfortable speed Walking (75% assistance): 4 min during back-and-forth locomotion on a 20-m length linear flat path, Trial 4 is not available in condition 1; Trial 5 - 1 minute Sit to stand test). Nasa TLX and RPE will be requested at the end of each trial. Usability questionnaires will be fullfilled at the end of condition 2 and condition 3.

SUMMARY:
The goal of this interventional study is to assess differences in the metabolic consumption, the cardiorespiratory effort, the cardiac autonomic adaptation, and fatigability during ADL, such as standing from a chair and walking while wearing an electrically powered exoskeleton in different modes of supports in subjects with neurological diseases with moderate to severe walking impairments.

DETAILED DESCRIPTION:
In people with severe gait impairments due to neurological diseases walk recovery is one primary goal, since achieving independent ambulation is a major contributing factor to their quality of life. Beyond walking, other very common Activities of Daily Living (ADL), such as postural transitions (which requires an integrity of the autonomic control mechanisms of blood pressure) and stair climbing (which requires the necessary strength in the lower limbs to lift one's own body weight) should be guaranteed by any rehabilitative intervention. Although physiotherapy treatments have proven effectiveness in improving gait and balance, conventional overground walking training may be very difficult or even impossible for patients with moderate to severe gait problems and limited cardiovascular capacity due to a too high energy demand (exercise intensity) (Calabrò 2022).

Wearable powered exoskeletons could be used to provide overground robotic assisted gait training (RAGT). Indeed, RAGT has shown clinically significant improvements in gait and balance outcomes and could be considered a valid approach to enhance gait function in people with severe gait impairments due to neurological diseases(Bowman 2021).

Little is known about the impact of robotic training on cardiovascular parameters and the metabolic / energy cost of walking with a wearable powered exoskeleton compared to unassisted overground walking in population with neurological diseases. It is possible that exoskeletons allow walking while keeping cardiorespiratory effort under control with a lower metabolic cost.

Moreover, people with severe gait impairments can suffer from disturbed cardiac autonomic control during exercise which affects exercise tolerance and balance during orthostatic challenges, such as the sit-to-stand maneuver. Indeed, to recommend RAGT in people with neurological diseases with moderate to severe gait impairments, the impact of the cardiac autonomic tone on sit-to-standing and walking with an exoskeleton should be investigated.

The use of an assisted as needed exoskeleton in clinical practice with population with moderate-severe neurological disabilities could increase their locomotor function by reducing the impact on metabolic consumption and cardiorespiratory effort compared to conventional overground walking training without an exoskeleton. Moreover, cardiovascular autonomic dysfunction (CAD), if any, should not be worsened by walking with an exoskeleton compared to conventional overground walking training, and should not constitute an impediment in the adaptation of the cardiovascular adaptation (especially of blood pressure) to the postural transitions.

The goal of this interventional study is to assess differences in the metabolic consumption, the cardiorespiratory effort, the cardiac autonomic adaptation, and fatigability during ADL, such as standing from a chair and walking while wearing an electrically powered exoskeleton in different modes of supports in subjects with neurological diseases with moderate to severe walking impairments.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform 4 minutes of back-and-forth locomotion with assistance or resting periods;
* Height between 160 and 195 cm;
* Weight not exceeding 100 kg;
* Diagnosis of Multiple Sclerosis with moderate to severe disability (5,5 < EDSS < 8,0);
* Diagnosis of stroke or traumatic brain damage (1 ≤ FAC ≤ 3);
* Diagnosis of spinal cord injury with neurological level of injury<T2 (3 ≤ WISCI II ≤ 16) with a Asia Impairment Score B, C or D.
* Able to perform 4 minutes of back-and-forth locomotion with assistance or resting periods;
* Able to use walker;

Exclusion Criteria:

* Impairments in the upper limbs that do not allow the user to hold the crutches/walker.
* Skin injuries in the areas where the exoskeleton is in contact with the user.
* Fractures not solved or bone pathologies in lower limbs in which the use of the exoskeleton could be risky (advanced osteoporosis).
* Psychiatric or cognitive problems that can interfere with the correct use of the device.
* Important muscle/joint retractions in lower limbs (Modified Ashworth Scale > 3).
* Any medical conditions that could interfere with the autonomic cardiovascular control (e.g severe diabetes).
* Use of beta blocker drugs.
* Presence of severe cardiovascular diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Walking meters change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  4 minutes walking test on a 20-meter corridor

SECONDARY OUTCOMES:
Number of repetitions change in one-minute sit to stand test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  The one-minute sit to stand test is performed with a chair of standard height without arm rests. The patient is ensured to be seated upright on the chair. The patient sat with the knees and hips flexed to 90°, feet placed flat on the floor hip-width apart, and the hands placed on the hips. Every get up from one's chair was validated to check if complete sit-to-stand-to-sit sequence was achieved.
Average VO2 change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Metabolic-related variables measured with K5-Cosmed device during 4 minute walking test on a 20-meter corridor
O2 cost of walking change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Metabolic-related variables measured with K5-Cosmed device during 4 minute walking test on a 20-meter corridor
Net metabolic power change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Metabolic-related variables measured with K5-Cosmed device during 4 minute walking test on a 20-meter corridor
Physiological cost index (PCI) change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Metabolic-related variables measured with PCI scale during 4 minute walking test on a 20-meter corridor
Average heart rate change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Cardiorespiratory parameters measured with pulse oximeter device during 4 minute walking test on a 20-meter corridor
Heart rate increase change during 4 minute walking test | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Cardiorespiratory parameters measured with pulse oximeter device during 4 minute walking test on a 20-meter corridor
Rating of perceived exertion of lower limbs change before and after each trials | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Fatigue-related parameters using the Borg scale scoring system ranging from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion".
Rating of perceived exertion of breath change before and after each trials | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Fatigue-related parameters using the Borg scale scoring system ranging from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion".
Assessment of device usability at the end of each condition | Baseline (Condition 2) and after 24 hours (Condition 3)
  Usability will be assessed with the System Usability Scale (SUS). SUS consists of a 10 item questionnaire with five response options for respondents; from "strongly agree" to "strongly disagree".
Assessment of users satisfaction at the end of each condition | Baseline (Condition 2) and after 24 hours (Condition 3)
  Satisfaction will be assessed with Telehealth satisfaction questionnaire (TSQWT). The TSQWT contains six subscales evaluating the benefit, usability, self-concept, privacy and loss of control, quality of life and wearing comfort of the system. Each subscale includes five questions rated on a 5-point Likert scale between 0 (I strongly disagree) and 4 (I strongly agree). The total score ranges between 0 (no satisfaction) and 120 (extreme satisfaction).
Assessment of the work load change during each trials | Baseline (Condition 1) and after 24 hours (Condition 2) and after 48 hours (Condition 3)
  Task load will be assessed with Nasa Task Load Index. NASA (TLX) method assesses work load on five 7-point scales. Increments of high, medium and low.

CONTACTS AND LOCATIONS:
Locations (4):
- Fondazione Don Carlo Gnocchi, Milan, MI, Italy
- Lithuanian University of Health Sciences, Kaunas, Lithuania
- Roessingh Research and Development, Enschede, AH, Netherlands
- Hospital Nacional de Parapléjicos de Toledo, Toledo, Spain